CLINICAL TRIAL: NCT00899756
Title: Study of Mutations of Epidermal Growth Factor Receptor in the Blood of Patients With Advanced Non Small Cell Lung Cancer
Brief Title: Epidermal Growth Factor Receptor Mutations in the Blood of Patients With Advanced Non-Small Cell Lung Cancer
Status: Completed | Type: Observational
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Other Study IDs: JS0538; CDR0000491609 (Registry Identifier: PDQ (Physician Data Query)); NA_00045719 (Other: JHM IRB)
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Molecular Diagnostic Techniques

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: molecular diagnostic method
Genetic: mutation analysis

SUMMARY:
RATIONALE: Collecting and storing samples of blood from patients with cancer to study in the laboratory may help doctors learn more about changes that may occur in DNA and identify biomarkers related to cancer.

PURPOSE: This laboratory study is looking at epidermal growth factor receptor mutations in the blood of patients with advanced non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine if epidermal growth factor receptor (EGFR) mutation exists in the peripheral blood of patients with advanced non-small cell lung cancer (NSCLC).
* Estimate the frequency of EGFR mutation in these patients.
* Correlate the presence of EGFR mutation in blood with EGFR mutation in primary or metastatic NSCLC tumor block.

OUTLINE: Patients undergo blood collection for analysis of epidermal growth factor receptor mutation by DNA sequencing.

PROJECTED ACCRUAL: A total of 50 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed advanced non-small cell lung cancer
* Must have available tumor tissue block

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any adult patient diagnosed with NSCLC with archiaved tissue availble.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2006-06 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Existence of epidermal growth factor receptor (EGFR) mutations in peripheral blood | Day 1
Frequency of EGFR mutation | Day 1
  Number of participants with EGFR mutation in tissue and plasma.
Number of participants with EGFR mutation in peripheral blood and in tumor tissue. | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Alex Y. Chang, MD, Study Chair — Johns Hopkins Singapore International Medical Centre
Locations (1):
- Alex Chang, Singapore, Singapore